CLINICAL TRIAL: NCT00164944
Title: Colonoscopic Screening in First-degree Relatives of Hong Kong Chinese Patients With Sporadic Colorectal Cancer: a Cohort Study With Case Control Analysis
Brief Title: Screening for Colorectal Neoplasm in First Degree Relatives of the Affected
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Other Study IDs: FDR
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer Screening
Keywords: Colonoscopy; First degree relatives
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FDR of CRC patient: First degree relatives of patients having CRC
  Interventions: Procedure: Colonoscopy
- FDR of normal colonoscopy: First degree relatives of patients having normal colonoscopy
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — To determine the adenomas during colonoscopy
  Groups: FDR of CRC patient
Procedure: Colonoscopy — To determine the adenomas during colonoscopy
  Groups: FDR of normal colonoscopy

SUMMARY:
To determine the prevalence of colorectal neoplasms in first degree relatives of those affected with sporadic colorectal cancer using colonoscopy as a screening tool. The prevalence will be compared to that of a defined matched cohort.

DETAILED DESCRIPTION:
Colorectal cancer is a second commonest tumor in Hong Kong and the second commonest cause of cancer related death. About 1 in 23 males will develop colorectal cancer in his life time. The disease tends to cluster in families. This may be a combination of factors including shared genes, shared environment or chance. Known familial syndromes occur in only about 5% of cases. The majority is not well understood and labelled sporadic colorectal cancer. The screening strategy in families of subjects with colorectal cancer has not been defined. Colonoscopy is among the most sensitive and specific screening tool for colorectal neoplasm. The current study determines the prevalence of adenomas among first degree relatives of patients diagnosed with colorectal cancer. To quantify risk in this cohort, a case control analysis is used. The prevalence of the cohort is compared to that of a control population. The control group consists of relatives of patients with normal colonoscopic findings during the same study period.

ELIGIBILITY:
Inclusion Criteria:

* First degree relatives (age >40 and <70) of individuals affected with sporadic colorectal cancer (those not associated with inflammatory bowel disease, familial adenomatous polyposis or HNPCC syndrome).

Exclusion Criteria:

* A family history compatible with that of Hereditary Non-polyposis Colon Cancer (HNPCC) based on the Amsterdam criteria [Table 5].
* Known Familial Adenomatous Polyposis (FAP) syndrome
* Patients and relatives with known inflammatory bowel disease
* Relatives that have received colonoscopy examinations in the past 5 years [details of colonoscopic examinations will be sought and information on colonic neoplasms recorded]. Those who have had barium enema examinations are eligible for trial inclusion as barium examinations often have low sensitivity and specificity for adenomas (around 70% respectively)
* Severe cardio-pulmonary or other medical co-morbidities that preclude safe colonoscopic examination

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First degree relatives of patients having CRC or patient having normal colonoscopy
Sampling Method: Probability Sample
Enrollment: 748 (Actual)
Dates: Start 2004-04; Primary Completion 2016-08 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
To find the prevalence of adenomas and advanced neoplasms of the first degree relatives | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: James Y Lau, MD, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong (sar), China

REFERENCES:
- [Derived] Ng SC, Lau JY, Chan FK, Suen BY, Leung WK, Tse YK, Ng SS, Lee JF, To KF, Wu JC, Sung JJ. Increased risk of advanced neoplasms among asymptomatic siblings of patients with colorectal cancer. Gastroenterology. 2013 Mar;144(3):544-50. doi: 10.1053/j.gastro.2012.11.011. Epub 2012 Nov 13. PMID 23159367